CLINICAL TRIAL: NCT06176768
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Efficacy and Safety of LY3972406 in Adults With Moderate-to-Severe Plaque Psoriasis
Brief Title: A Study of LY3972406 in Adult Participants With Moderate-to-Severe Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18692; J4H-MC-FVAA (Other: Eli Lilly and Company); 2023-504485-39-00 (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3972406 (Experimental): Participants received an oral dose of LY3972406 for 12 weeks.
  Interventions: Drug: LY3972406
- Placebo (Placebo Comparator): Participants received an oral dose of placebo for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3972406 — Administered orally
  Arms: LY3972406
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The main purpose of this study is to determine the efficacy and safety of LY3972406 in adult participants with moderate-to-severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Have moderate-to-severe chronic plaque psoriasis for at least 6 months prior to baseline
* Have venous access sufficient to allow for blood sampling
* Are able to swallow oral medication

Exclusion Criteria:

* Have any other skin conditions, excluding plaque psoriasis
* Have a current or recent acute, active infection
* Have manifestations of other autoimmune diseases, such as systemic lupus erythematosus.
* Are lactating or breastfeeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-12-06 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 on - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (12):
- United States (12):
  - Dermatology Research Associates, Los Angeles, California
  - Clinical Science Institute, Santa Monica, California
  - Driven Research, Coral Gables, Florida
  - Conquest Research, Winter Park, Florida
  - Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - Schweiger Dermatology Group, Hackensack, New Jersey
  - Metropolitan Dermatology - Clark, Kenilworth, New Jersey
  - Accellacare - Winston-Salem, Winston-Salem, North Carolina
  - Remington-Davis, Inc, Columbus, Ohio
  - DermDox Centers for Dermatology, Camp Hill, Pennsylvania
  - Center for Clinical Studies, Houston, Texas
  - Austin Institute for Clinical Research, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LY3972406 | Placebo
Started | 16 | 17
Received at Least 1 Dose of the Study Drug | 16 | 17
Completed | 3 | 4
Not Completed | 13 | 13
Not completed — Adverse Event | 1 | 0
Not completed — Assigned treatment by mistake | 1 | 0
Not completed — Lost to Follow-up | 0 | 3
Not completed — Physician Decision | 1 | 0
Not completed — Protocol deviation | 3 | 1
Not completed — Other | 1 | 0
Not completed — Withdrawal by Subject | 6 | 9

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | LY3972406 | Placebo | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (13.3) | 50.2 (13.5) | 50.3 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 15 | 14 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 10 | 23
  Not Hispanic or Latino | 3 | 7 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 12 | 11 | 23
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving ≥75% Reduction From Baseline in Psoriasis Area and Severity Index (PASI-75)
Description: * The PASI is an investigator-administered, multi-item scale used to measure the severity of psoriasis based on lesion severity and the percent of body surface area (BSA) affected.
  * Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomical regions: head, trunk, upper limbs, lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement).
  * The sum of severity scores for erythema, thickness, and scaling is multiplied by the degree of involvement for each anatomic region, and then multiplied by a constant corresponding to the region's percent BSA (0.1, 0.3, 0.2, and 0.4 for the above 4 regions, respectively). The resultant score for each anatomic region is then summed to yield the final PASI score. It ranges from 0 to 72, with higher scores reflecting greater disease severity.
  * The nonresponder imputation (NRI) method was used to handle missing data.
Time Frame: Week 12
Population: All randomized participants who received at least one dose of the study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LY3972406 | Placebo
Number analyzed (Participants) | 16 | 17
percentage of participants | 18.8 [0 to 37.9] | 5.9 [0 to 17.1]
Statistical Analysis 1: Comparison: LY3972406 vs Placebo; Test type: Superiority; p = 0.316, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.4, 95% CI 2-sided [0.3 to 40.4]

2. Secondary Outcome: Change From Baseline in Percent Body Surface Area (BSA)
Description: The percent BSA is the total percentage of psoriasis involvement on the participant's body surface, ranging from 0% (no involvement) to 100% (full involvement). It is measured using the handprint method, where 1% corresponds to the size of the participant's hand (including the palm, fingers, and thumb). The number of handprints fitting into the affected areas across the body is summed to estimate the total percentage of involvement.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of the study drug and had non-missing values for this outcome at week 12.
Measure: Least Squares Mean (Standard Error); unit: percent BSA
Arm/Group | LY3972406 | Placebo
Number analyzed (Participants) | 11 | 10
percent BSA | -7.26 (3.35) | -0.48 (3.19)
Statistical Analysis 1: Comparison: LY3972406 vs Placebo; Test type: Superiority; p = 0.175, Mixed Model Repeated Measures Analysis; Least square mean difference = -6.77, 95% CI 2-sided [-17.15 to 3.60], Standard Error of Mean 4.63

3. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI)
Description: The DLQI is a validated, dermatology-specific, patient-reported outcomes 10-item questionnaire that evaluates participants health-related quality of life over the past week. The 10 questions are grouped into 6 domains, including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. Response categories and corresponding scores are:
  * Very much = 3
  * A lot = 2
  * A little = 1
  * Not at all = 0
  * Not relevant = 0.
  The total score is calculated by summing all 10 question responses and has a range of 0 (no impact of skin disease on quality of life) to 30 (maximum impact on quality of life).
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | LY3972406 | Placebo
Number analyzed (Participants) | 11 | 11
score on a scale | -6.71 (1.64) | -4.35 (1.54)
Statistical Analysis 1: Comparison: LY3972406 vs Placebo; Test type: Superiority; p = 0.311, Mixed Model Repeated Measures Analysis; Least square mean difference = -2.36, 95% CI 2-sided [-7.06 to 2.35], Standard Error of Mean 2.27

4. Secondary Outcome: Pharmacokinetics (PK): Observed Trough Plasma Concentration of LY3972406
Description: Observed trough plasma concentration (Ctrough) of LY3972406.
Time Frame: Predose at Week 12
Population: All randomized participants who received at least one dose of the study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | LY3972406
Number analyzed (Participants) | 8
Nanogram per milliliter (ng/mL) | 158 (155)

ADVERSE EVENTS:
Time Frame: From baseline to the end of follow-up (up to Week 24)
Description: All randomized participants who received at least 1 dose of the study drug.
Arm/Group | LY3972406 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/16 | 1/17
Other Adverse Events (participants affected / at risk) | 9/16 | 6/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY3972406 (N=16) | Placebo (N=17)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY3972406 (N=16) | Placebo (N=17)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Eczema eyelids (Eye disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2024-07-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT06176768/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-02): https://cdn.clinicaltrials.gov/large-docs/68/NCT06176768/SAP_001.pdf